CLINICAL TRIAL: NCT03015285
Title: Comparing the Efficacy of CBT for Anxiety Sensitivity to Disorder-specific CBT in Reducing Mental Health Symptoms: A Randomized Controlled Trial
Brief Title: CBT for Anxiety Sensitivity vs. Disorder-specific CBT: An RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: University of New Brunswick (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1021903
Record Dates: First submitted 2016-12-19; First posted 2017-01-10 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Generalized Anxiety; Stress Disorder, Posttraumatic; Social Anxiety; Major Depression; Panic Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anxiety Sensitivity Cognitive Therapy (Experimental): Participants in the Cognitive Behavioural Therapy for AS condition will complete 8 weekly 50-minute therapy sessions and will be asked to continue with some parts of the intervention (i.e., interoceptive exposure) independently for the next 4 weeks, with short weekly check-ins by phone with their therapist.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Disorder specific Cognitive Therapy (Active Comparator): Participants in the disorder-specific Cognitive Behavioural Therapy intervention will receive 12 weekly 50-minute therapy sessions following established, evidence-based protocols for each of the disorders included in the study.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — A type of talk therapy called cognitive behaviour therapy (CBT) will be delivered to both groups.

SUMMARY:
Adults with high anxiety sensitivity (AS) and a mental health diagnosis of anxiety, depression, or posttraumatic stress will be recruited and will be randomly assigned to either transdiagnostic cognitive behavioural therapy (CBT) for AS or disorder-specific CBT for their primary mental health problem. The study outcomes - AS, anxiety, mood, and substance use symptoms, and functional impairment - will be assessed at pre-and post-treatment and 6 and 12 months post-treatment via standardized self-report measures completed by participants and a standardized diagnostic interview.

DETAILED DESCRIPTION:
While our previous work has provided some evidence that cognitive behavioural therapy (CBT) for anxiety sensitivity(AS) reduces mental health symptoms, the current study aims to determine whether this treatment works as well as traditional disorder-specific CBT (which aims to treat the specific disorder a person presents with, such as CBT for panic disorder for someone with panic disorder) in treating anxiety and depression. This will be the first study to have looked at this question.

Our objectives are to determine:

1. if there is a difference in the extent to which CBT for AS vs. disorder-specific CBT reduces, in the short- and long-term, a) AS, b) symptoms of a person's primary and secondary mental health problems, and c) functional disability (i.e., a person's ability to function in day-to-day life);
2. if the two treatments lead to differences in the number of participants who no longer meet the requirements for a diagnosis (of their primary or secondary mental health problems) in the short- and long-term; and
3. if the treatments are seen as similarly satisfactory by participants.

Eligible participants will be randomly assigned (via online random number generator) to either transdiagnostic CBT for AS or disorder-specific CBT for their primary mental health problem. Both CBT interventions are evidence-based, guided by treatment manuals/workbooks (provided to participants), and involve 12 weekly therapy sessions. The AS intervention will also involve a physical exercise component (i.e., running/brisk walking 3x/week starting on week 5) and participants will be provided with a wearable fitness device designed to provide physiological indices of arousal and track physical activity. The study outcomes - AS, anxiety, mood, and substance use symptoms, and functional impairment - will be assessed at pre-and post-treatment and 6 and 12 months post-treatment via standardized self-report measures completed by participants and a standardized diagnostic interview.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* High Anxiety Sensitivity (high AS, participants must score ≥23 on the Anxiety Sensitivity Index - 3)
* Live in the surrounding area of Halifax, Nova Scotia or Fredericton, New Brunswick
* Must have a primary diagnosis of one of Agoraphobia, Generalized Anxiety Disorder (GAD), Social Anxiety Disorder (SAD), Panic Disorder (PD), Other Specified Anxiety Disorder, Major Depressive Disorder (MDD), Posttraumatic Stress Disorder (PTSD), or Illness Anxiety Disorder (IAD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5; APA, 2013) as determined by a Structured Clinical Interview for DSM-5 Disorders

Exclusion Criteria:

* Must not have any contraindications to physical exercise
* Must not be engaged in another current psychotherapy as it may interfere with the treatment under investigation
* Need to be able to attend intervention sessions at Dalhousie University or the University of New Brunswick
* Must not have current Bipolar Disorder and psychosis nor current suicidal intent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Change in anxiety sensitivity: the Anxiety Sensitivity Index - 3 (ASI-3) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up.
  The ASI-3 is an 18-item self-report measure that indexes the amount of fear an individual experiences with respect to anxiety-related body sensations. Participants indicate the extent to which they agree or disagree with each item (e.g., "It scares me when my heart beats rapidly") on a 5-point Likert-type scale.
Change in primary diagnosis (e.g., anxiety disorder or depression) symptoms | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  Primary diagnosis (e.g., anxiety disorder or depression) symptoms, as measured by a standardized score on one of the Panic Attack Questionnaire - IV, the Fear Questionnaire, the Generalized Anxiety Disorder - 7-item, the Liebowitz Social Anxiety Scale, the PTSD Checklist for DSM-5, the Pain Anxiety Symptom Scale - 20-item, or the Patient Health Questionnaire - 9-item.
Change in comorbid diagnosis (e.g., anxiety disorders or depression) symptoms | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up.
  Comorbid diagnosis (e.g., anxiety disorder or depression) symptoms, as measured by a standardized score on one of the Panic Attack Questionnaire - IV, the Fear Questionnaire, the Generalized Anxiety Disorder - 7-item, the Liebowitz Social Anxiety Scale, the PTSD Checklist for DSM-5, the Pain Anxiety Symptom Scale - 20-item, or the Patient Health Questionnaire - 9-item.

SECONDARY OUTCOMES:
Diagnostic status as measured by the Structured Clinical Interview for DSM-5 (SCID-5) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  Administered by a trained researcher blind to treatment condition. The SCID-5 has been widely used in numerous research studies and is well empirically validated. At each time point, we will assess participants' primary and secondary diagnoses as well as the overall number of diagnoses for which they qualify.
General distress as measured by the Depression Anxiety Stress Scale (DASS-21) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  The Depression Anxiety Stress Scales - 21. The DASS-21 is a shortened version of the 42-item DASS and is composed of three subscales: Depression, Anxiety, and Stress. Individuals indicate the extent to which a particular negative emotional state (e.g., "I found it difficult to relax") has applied to them over the past week on a 4-point Likert-type scale (0 = Did not apply to me at all to 3 = Applied to me very much or most of the time).
General distress as measured by the Clinical Outcomes in Routine Evaluation measure (CORE-10) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  Clinical Outcomes in Routine Evaluation (CORE-10) is a brief, 10-item self-report measure designed to assess common presentations of symptoms of psychological distress. Participants are asked to indicate how often in the past week they have felt a series of symptoms (e.g., "I have felt tense, anxious, or nervous") on a 5-point Likert-type scale.
Functional disability as measured by the Sheehan Disability Scale (SDS) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  The Sheehan Disability Scale will be used to measure functional impairment in three domains: work/school, family life, and social. Using a 10-point visual analogue scale, participants rate the extent to which their general mental health symptoms disrupt their work/school, family life/responsibilities, and social life. Participants also indicate the number of days their mental health symptoms caused them to miss school/work as well as the number of days their symptoms had caused their performance to be reduced during the past week. The SDS is well-validated and widely used with a range of populations.
Drinking Motives as measured by the Modified Drinking Motives Questionnaire - Revised (MDMQ-R) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  The MDMQ-R measures drinking motives. Respondents estimate how often they drink for the reason specified in each item on a 5-point Likert-type scale.
Hazardous alcohol use as measured by the Alcohol Use Disorders Identification Test (AUDIT) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  Despite being designed as a screening tool, the AUDIT is commonly used to assess alcohol use problems pre- and post-treatment. The AUDIT is a 10-item self-report measure that asks participants to report on their frequency of alcohol use, binge drinking, and alcohol-dependent behaviours. Responses are scored on 5-point Likert-type scales. Finally, participants report if they have experienced problems caused by alcohol use on a 3-point Likert-type scale.
Alcohol-related problems as measured by the Short Inventory of Problems (SIP-2R) | baseline (i.e., start of study), 12 weeks, 6 months, and 12 months follow-up
  The SIP-2R consists of the three items from each of five subscales. Participants are asked to indicate the frequency with which they have experienced each of 15 drinking-related problems on a 4-point Likert-type scale.
Treatment alliance as measured by the Working Alliance Inventory - Short-form (WAI-SR) | Only at 12 weeks
  The WAI-SR is a 12-item self-report questionnaire comprised of three subscales: Goals, or agreement on the goals of therapy, Tasks, or agreement on the tasks of therapy, and Bonds, or the bond between the therapist and the client. Participants indicate the extent to which each of these statements reflects their experience on a 5-point Likert-type scale.
Treatment satisfaction as measured by several short researcher-generated questions | Only at 12 weeks
  In order to assess satisfaction with the different components of treatment, participants will answer a series of open-ended questions about their experience (e.g., "Was the treatment convenient for you to engage in?"; "Did you find the telephone therapy sessions helpful?") after all parts of treatment are completed (i.e., at 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Margo Watt, PhD, Principal Investigator — St. Francis Xavier University; Janine Olthuis, PhD, Principal Investigator — University of New Brunswick

IPD SHARING:
Plan to Share IPD: No
Data will only be shared between investigators at the two study sites once it has been de-identified and entered into a data analytic program in order to protect participants' privacy and confidentiality.